CLINICAL TRIAL: NCT05316428
Title: A Randomized, Blind, Placebo-controlled, Three-way Crossover Study Evaluating the Interaction of TPN171H Tablets and Alcohol in Healthy Chinese Male Subjects
Brief Title: A Study of the Hemodynamic Interactions of TPN171H Tablets & Alcohol in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vigonvita Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TPN171H-08
Record Dates: First submitted 2022-02-08; First posted 2022-04-07 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-02

CONDITIONS: Alcohol; Phosphodiesterase Inhibitor; Erectile Dysfunction
Keywords: Phase I; Crossover Study; Alcohol; TPN171H
MeSH Terms: conditions — Erectile Dysfunction | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- alcohol plus TPN171H (Experimental): 0.5 g/Kg alcohol plus 10 mg TPN171H tablet
  Interventions: Drug: TPN171H tablet plus alcohol
- alcohol (Experimental): 0.5 g/kg alcohol
  Interventions: Other: alcohol
- TPN171H (Experimental): 10 mg TPN171H tablet
  Interventions: Drug: TPN171H tablet

INTERVENTIONS:
Drug: TPN171H tablet plus alcohol — 10 mg TPN171H tablet QD plus 0.5 g/kg alcohol
  Arms: alcohol plus TPN171H
Other: alcohol — 0.5 g/kg alcohol
  Arms: alcohol
Drug: TPN171H tablet — 10 mg TPN171H tablet QD
  Arms: TPN171H

SUMMARY:
The purpose of this study is primarily to evaluate the effects of taking TPN171H tablets with alcohol on blood pressure, pulse,and pharmacokinetic in Chinese healthy male subjects.

DETAILED DESCRIPTION:
This study will be divided into two parts: pre-test and formal test. The pre-trial is an open design to evaluate the safety and tolerability of TPN171H tablets in combination with alcohol in healthy male subjects. Two subjects at 5 mg and 10 mg doses will be taken with alcohol, blood pressure (SBP and DBP), pulse, alcohol breath monitoring and PK blood sample collection were required, and the time point was the same as the formal test.

The dosage of TPN171H tablets in the formal trial will be determined according to the preliminary test results.

The formal trial is a single-centre, blind, randomized, placebo-controlled, three-period, three-way crossover study, in which each subject will be randomized to receive each of the following three treatments with a washout period of at least 3 days between treatments:

Treatment A: a single oral dose of one10 mg or 5 mg TPN171H tablet plus an oral dose of alcohol drink mixed with fruit juice (0.5 g of absolute ethanol per kilogram of body weight).

Treatment B: a single oral dose of one placebo tablet plus an oral dose of alcohol drink mixed with fruit juice (0.5 g of absolute ethanol per kilogram of body weight).

Treatment C: a single oral dose of one10 mg or 5 mg TPN171H tablet plus an oral dose of placebo drink mixed with fruit juice.

For each treatment period, supine blood pressure and pulse rate will be measured pre-dose and every 15 minutes for 4 hours post-dose,and at 6h,8h,24h and 48h post-dose. Alcohol levels using a breathalyzer will be measured at pre-dose and up to 8 hours post dose during all 3 treatments by designated unblinded personnel.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign and abide by the contents of the informed consent;
2. Adult male subjects, either 21 to 45 years of age,
3. Body weight ≥55 kg; Body mass index (BMI) in the range of 19.0-26.0 kg/m2 (including the critical value);
4. Subjects must agree to use at least one method of birth control for at least three months from the time of the first dose to at least the last;
5. Normal or abnormal important indicators of physical examination, vital signs examination, electrocardiogram examination and laboratory examination have no clinical significance as judged by the researcher.

Exclusion Criteria:

1. Unable to consume alcohol according to 0.5 g/kg (body weight);
2. After ingestion of 0.5 g/kg alcohol, the instrument showed alcohol concentration ≥120 mg/100 mL after exhalation, or moderate or severe acute alcoholism, which was judged by the investigator to be unfit to continue to participate in the study (see Appendix 1 for clinical classification of acute alcoholism);
3. Systolic pressure in decubitus (semi-decubitus) position < 90 or ≥140 mmHg; Diastolic pressure in decubitus (semi-decubitus) position < 60 or ≥90 mmHg；
4. Known allergic history, patients with allergic diseases or allergic predisposition to the study product or any of its components or related product;
5. May significantly affect drug absorption, distribution, metabolism and excretion of any surgical situation or condition, or may pose a hazard to participate in research subjects of any surgical situation or condition, such as the history of gastrointestinal surgery (gastrectomy, gastrointestinal anastomosis, intestinal resection, etc.), gastroenteritis, gastrointestinal ulcers, gastrointestinal bleeding history etc. (except for gallbladder removal);
6. Patients with myocardial infarction, severe/unstable angina pectoris, coronary artery/peripheral artery bypass graft, congestive heart failure, severe arrhythmias, and cerebrovascular accidents, including transient ischemic attack, within 6 months prior to the administration of the study drug;
7. Those who had used any drugs to inhibit or induce drug metabolism in the liver within 4 weeks before enrollment or needed to use any drugs in combination during the study period; Patients taking nitrates in any form;
8. Known history of the following eye diseases: non-avascular ischemic optic neuropathy (NAION), abnormal color vision, hereditary retinal degeneration (e.g. Retinitis pigmentosa), macular degeneration;
9. Known history of sudden hearing loss or loss;
10. A history of postural hypotension;
11. Patients with blood loss >400 mL within 3 months before inclusion;
12. Participated in clinical research of other drugs or medical devices within 3 months prior to inclusion;
13. Current or previous alcoholics (drinking more than 14 standard units per week. 1 standard unit containing 14 g alcohol, such as 360 mL beer or 45 mL 40% spirits or 150 mL wine), or positive breath test for alcohol;
14. Have a history of drug use or have been screened positive for drug abuse;
15. Smokers who smoked more than 10 cigarettes a day within 6 months prior to inclusion;
16. Human immunodeficiency virus antibody (HIV), hepatitis C virus antibody (anti-HCV), hepatitis B surface antigen (HBsAg), treponema pallidum antibody (anti-TP) positive;
17. Alcohol sensitivity test positive;
18. There were other factors that the investigator considered inappropriate for the study.

Ages: 21 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2022-04-02 (Actual); Study Completion 2022-04-06 (Actual)

PRIMARY OUTCOMES:
Maximum change in blood pressure (SBP and DBP) | 48 hours after treatment
  Maximum change in decubitus (semi-decubitus) blood pressure (SBP and DBP) from baseline
Maximum change in pulse | 48 hours after treatment
  Maximum change from baseline in decubitus (semi-decubitus) position;
The area under effect-time curve (AUEC0- 4h) of supine systolic (SBP) and diastolic (DBP) blood pressure, and pulse | 4 hours after treatment
  The area under effect-time curve (AUEC0- 4h) of supine systolic (SBP) and diastolic (DBP) blood pressure, and pulse relative to baseline change.

CONTACTS AND LOCATIONS:
Overall Officials: Chen Yu, Principal Investigator — Shanghai Xuhui Central Hospital
Locations (1):
- Shanghai Xuhui Central Hospital, Shanghai, China